CLINICAL TRIAL: NCT02474329
Title: Real-PD: Development of Clinical Prognostic Models for Parkinson's Disease From Large-scale Wearable Sensor Deployment and Clinical Data - a Population Based Trial
Brief Title: Real-PD Trial: Development of Clinical Prognostic Models for Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other); Philips Electronics Nederland B.V. acting through Philips CTO organization (Industry); Intel Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: NL53034.091.41
Record Dates: First submitted 2015-06-02; First posted 2015-06-17 (Estimated); Results first posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2017-10

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Ambulatory monitoring; Disease progression
MeSH Terms: conditions — Parkinson Disease; Disease Progression | interventions — Clinical Protocols

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 13 Weeks
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Cohort 1: Dutch Parkinson's patients resident in the region of Noord-Holland whose fulfill the eligibility criteria.
  Interventions/Exposures to be administered:
  1. PPMI (Parkinson's Progression Markers Initiative) protocol Trained physiotherapists will perform once a standardized clinical assessment to every included patient. This assessment will last for 60 minutes, and it will be done once.
  2. Fox Insight self-monitoring android app and falls detector Patients will wear a smartwatch and a pendant movement sensor during day and night, for a period of 13 weeks. Additionally, a self-monitoring App on a Smartphone is used, where the patient reports when (s)he takes any PD medication. An additional, optional button allows the patient to report general feeling.
  Interventions: Other: Clinical assessment; Device: Fox Insight self-monitoring android app and falls detector
- Cohort 2: Dutch Parkinson's patients resident in the region of Zuid-Holland whose fulfill the eligibility criteria.
  Interventions/Exposures to be administered:
  1. PPMI (Parkinson's Progression Markers Initiative) protocol Trained physiotherapists will perform once a standardized clinical assessment to every included patient. This assessment will last for 60 minutes, and it will be done once.
  2. Fox Insight self-monitoring android app and falls detector Patients will wear a smartwatch and a pendant movement sensor during day and night, for a period of 13 weeks. Additionally, a self-monitoring App on a Smartphone is used, where the patient reports when (s)he takes any PD medication. An additional, optional button allows the patient to report general feeling.
  Interventions: Other: Clinical assessment; Device: Fox Insight self-monitoring android app and falls detector
- Cohort 3: Dutch Parkinson's patients resident in the region of Gelderland and Utrecht whose fulfill the eligibility criteria.
  Interventions/Exposures to be administered:
  1. PPMI (Parkinson's Progression Markers Initiative) protocol Trained physiotherapists will perform once a standardized clinical assessment to every included patient. This assessment will last for 60 minutes, and it will be done once.
  2. Fox Insight self-monitoring android app and falls detector Patients will wear a smartwatch and a pendant movement sensor during day and night, for a period of 13 weeks. Additionally, a self-monitoring App on a Smartphone is used, where the patient reports when (s)he takes any PD medication. An additional, optional button allows the patient to report general feeling.
  Interventions: Other: Clinical assessment; Device: Fox Insight self-monitoring android app and falls detector
- Cohort 4: Dutch Parkinson's patients resident in the region of Groningen, Friesland, Drenthe and Overijssel whose fulfill the eligibility criteria.
  Interventions/Exposures to be administered:
  1. PPMI (Parkinson's Progression Markers Initiative) protocol Trained physiotherapists will perform once a standardized clinical assessment to every included patient. This assessment will last for 60 minutes, and it will be done once.
  2. Fox Insight self-monitoring android app and falls detector Patients will wear a smartwatch and a pendant movement sensor during day and night, for a period of 13 weeks. Additionally, a self-monitoring App on a Smartphone is used, where the patient reports when (s)he takes any PD medication. An additional, optional button allows the patient to report general feeling.
  Interventions: Other: Clinical assessment; Device: Fox Insight self-monitoring android app and falls detector
- Cohort 5: Dutch Parkinson's patients resident in the region of Zeeland, Noord-Brabant and Limburg whose fulfill the eligibility criteria.
  Interventions/Exposures to be administered:
  1. PPMI (Parkinson's Progression Markers Initiative) protocol Trained physiotherapists will perform once a standardized clinical assessment to every included patient. This assessment will last for 60 minutes, and it will be done once.
  2. Fox Insight self-monitoring android app and falls detector Patients will wear a smartwatch and a pendant movement sensor during day and night, for a period of 13 weeks. Additionally, a self-monitoring App on a Smartphone is used, where the patient reports when (s)he takes any PD medication. An additional, optional button allows the patient to report general feeling.
  Interventions: Other: Clinical assessment; Device: Fox Insight self-monitoring android app and falls detector

INTERVENTIONS:
Other: Clinical assessment — During the 13 week follow-up, trained physiotherapists will perform a standardized clinical assessment, based on the PPMI protocol (www.ppmi-info.org) for every included patient. This assessment will last for 60 minutes, and it will be done once.
  Other Names: PPMI (Parkinson's Progression Markers Initiative) protocol
Device: Fox Insight self-monitoring android app and falls detector — Patients will be asked to wear a smartwatch and a pendant movement sensor, both with triaxial accelerometers, during day and night, for a period of 13 weeks. Additionally, a self-monitoring App on a Smartphone is used, where the patient reports when (s)he takes any PD medication. An additional, optional button allows the patient to report general feeling.
  Other Names: Pebble smartphone; Philips falls detector

SUMMARY:
Background: Long-term management of Parkinson's disease (PD) does not reach its full potential due to lack of knowledge about disease progression. The Real-PD study aim to evaluate the feasibility and compliance of usage of wearable sensors in PD patients in real life. Moreover, an explorative analysis concerning activity level, medication intake and mood will be done.

Methods: Overall, 1000 PD patients and 250 physiotherapist will be enrolled in this observational study. Dutch PD patients will be recruited across the country and an assessment will be performed using a short version of the Parkinson's Progression Markers Initiative (PPMI) protocol. Moreover, participants will wear a set of medical devices (Pebble Smartwatch, fall detector) and they will use a smartphone with The Fox Insight App (Android app), 24/7, during 13 weeks. Primary measures of interest are: 1) physical activity, falls and tremor, measured by the axial accelerometers embedded in the Pebble watch and fall detector; and 2) medication intake and mood reports measured by patients' self-report in the Android app. To measure motor impact, an assessment will be performed by physiotherapists who are all certified to perform the Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS).

Discussion: Management of PD patients is complex and appears to be a challenging task for health care professionals. The main reason is the lack of knowledge in the disease pattern. This issue could be solved by a long term follow-up of patients' during their everyday life, and wearable medical devices can act as a way to collect data about every day life activities. Therefore, the Real-PD study will be a first contribution in increasing the lack of knowledge in disease progression, developing a new medical decision system and improving PD patients' care.

DETAILED DESCRIPTION:
Rationale: Today's management of patients with a chronic disorder like Parkinson's disease (PD) is imperfect. The understanding of clinical profiles is based on observations in small, selective populations with brief follow-up. Moreover, treatment decisions are based on averaged population results that may not apply to a specific individual context. These drawbacks will be addressed with a "big data" approach. Ambulatory sensors will be used as an objective measure of patients' performance under everyday circumstances, for longer periods of time. The researchers aim to explore the potential of using longitudinal ambulatory data to enrich a standardized clinical dataset, which reflects current clinical practice for the assessment of disease status.

Objective: The study will include a total of 250 physiotherapists and 1000 patients. The aims of this study are: (1) to perform "big data" analyses on the raw sensor data, in relation to concurrently acquired clinical data in these patients (limited version of the PPMI (Parkinson's Progression Markers Initiative) protocol) to develop patient profiles; and (2) to correlate the ambulatory sensor data to simple self-assessments made during follow-up.

Study design: Observational descriptive study.

Study population: Dutch Parkinson patients, male or female, age 30 years or older, with PD diagnosis given by a physician, and own a suitable smartphone.

lntervention: 250 ParkinsonNet physiotherapists and 1000 eligible patients will be included in this study. Patients and physiotherapists will be recruited in 5 consecutive cohorts based on geographic region. Patients will be asked to wear a smartwatch and a pendant movement sensor, both with triaxial accelerometers, during day and night, for a period of 13 weeks. Additionally, a self-monitoring App on a smartphone is used, where the patient reports when (s)he takes any PD medication. An additional, optional button allows the patient to report general feeling. During the 13 week follow-up, trained physiotherapists will perform a standardized clinical assessment, based on the PPMI protocol (www.ppmi-info.org) for every included patient. This assessment will last for 60 minutes. The smartphone is used to transmit data from the watch to a cloud-based data platform. lntel developed this dedicated data analysis platform for ambulatory data. lntel will receive coded data only.

Main study parameters/endpoints: Study endpoints include parameters registered with the smartwatch, the pendant movement sensor, the self-monitoring app and collected with the PPMI assessment. The smartwatch data provides, after data processing, a measure for the level of physical activity during the day. Falls will be registered with the pendant movement sensor. Medication intake and mood are registered using the smartphone. Finally, PPMI assessment includes assessment of motor symptoms, cognition, depression, sleep and daily activity. Correlations will be determined between the above mentioned parameters.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: First, participants are asked to wear the devices 24/7 and data will be recorded continuously, for a total duration of 13 weeks. Second, data will be transmitted to a data platform developed and managed by lntel, on behalf of the Michael J. Fox Foundation for Parkinson's Research. To access these data, researchers can grant permission for research purposes, provided by Michael J. Fox Foundation. Patients will be asked for permission to share the raw coded data for dissemination to the research community, analysis and use in future publications. Participation in the study warrants that patients provide written permission for this.

ELIGIBILITY:
Inclusion Criteria:

1. Currently own and use a smartphone device with access to the Internet
2. 30 years of age or older;
3. Diagnosed with Parkinson's disease by a physician;
4. Able to walk without any assistance.

Exclusion Criteria:

None exclusion criteria will be used.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dutch Parkinson patients.
Sampling Method: Non-Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2015-07; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bastiaan R Bloem, Prof. Dr., Principal Investigator — Radboud University Medical Center
Locations (1):
- Cohort 1, Multiple Locations, North Holland, Netherlands

REFERENCES:
- [Background] Parkka J, Ermes M, Korpipaa P, Mantyjarvi J, Peltola J, Korhonen I. Activity classification using realistic data from wearable sensors. IEEE Trans Inf Technol Biomed. 2006 Jan;10(1):119-28. doi: 10.1109/titb.2005.856863. PMID 16445257
- [Background] Hobert MA, Maetzler W, Aminian K, Chiari L. Technical and clinical view on ambulatory assessment in Parkinson's disease. Acta Neurol Scand. 2014 Sep;130(3):139-47. doi: 10.1111/ane.12248. Epub 2014 Apr 1. PMID 24689772
- [Background] Maetzler W, Domingos J, Srulijes K, Ferreira JJ, Bloem BR. Quantitative wearable sensors for objective assessment of Parkinson's disease. Mov Disord. 2013 Oct;28(12):1628-37. doi: 10.1002/mds.25628. Epub 2013 Sep 12. PMID 24030855
- [Background] Patel S, Lorincz K, Hughes R, Huggins N, Growdon J, Standaert D, Akay M, Dy J, Welsh M, Bonato P. Monitoring motor fluctuations in patients with Parkinson's disease using wearable sensors. IEEE Trans Inf Technol Biomed. 2009 Nov;13(6):864-73. doi: 10.1109/TITB.2009.2033471. Epub 2009 Oct 20. PMID 19846382
- [Background] Patel S, Chen BR, Mancinelli C, Paganoni S, Shih L, Welsh M, Dy J, Bonato P. Longitudinal monitoring of patients with Parkinson's disease via wearable sensor technology in the home setting. Annu Int Conf IEEE Eng Med Biol Soc. 2011;2011:1552-5. doi: 10.1109/IEMBS.2011.6090452. PMID 22254617
- [Background] Tsanas A, Little MA, McSharry PE, Ramig L. Using the cellular mobile telephone network to remotely monitor parkinsons disease symptom severity. IEEE Transactions on Biomedical Engineering. 2012.
- [Background] Arora S, Venkataraman V, Donohue S, Biglan KM, Dorsey ER, Little MA, editors. High accuracy discrimination of Parkinson's disease participants from healthy controls using smartphones. Acoustics, Speech and Signal Processing (ICASSP), 2014 IEEE International Conference on; 2014: IEEE.
- [Background] Pastorino M, Arredondo M, Cancela J, Guillen S, editors. Wearable sensor network for health monitoring: the case of Parkinson disease. Journal of Physics: Conference Series; 2013: IOP Publishing.
- [Background] Sharma V, Mankodiya K, De La Torre F, Zhang A, Ryan N, Ton TG, et al. SPARK: Personalized Parkinson Disease Interventions through Synergy between a Smartphone and a Smartwatch. Design, User Experience, and Usability User Experience Design for Everyday Life Applications and Services: Springer; 2014. p. 103-14.
- [Background] Tzallas AT, Tsipouras MG, Rigas G, Tsalikakis DG, Karvounis EC, Chondrogiorgi M, Psomadellis F, Cancela J, Pastorino M, Waldmeyer MT, Konitsiotis S, Fotiadis DI. PERFORM: a system for monitoring, assessment and management of patients with Parkinson's disease. Sensors (Basel). 2014 Nov 11;14(11):21329-57. doi: 10.3390/s141121329. PMID 25393786
- [Background] Lakshminarayana R, Wang D, Burn D, Chaudhuri KR, Cummins G, Galtrey C, Hellman B, Pal S, Stamford J, Steiger M, Williams A; SMART-PD Investigators. Smartphone- and internet-assisted self-management and adherence tools to manage Parkinson's disease (SMART-PD): study protocol for a randomised controlled trial (v7; 15 August 2014). Trials. 2014 Sep 25;15:374. doi: 10.1186/1745-6215-15-374. PMID 25257518
- [Background] Gschwind YJ, Eichberg S, Marston HR, Ejupi A, Rosario Hd, Kroll M, Drobics M, Annegarn J, Wieching R, Lord SR, Aal K, Delbaere K. ICT-based system to predict and prevent falls (iStoppFalls): study protocol for an international multicenter randomized controlled trial. BMC Geriatr. 2014 Aug 20;14:91. doi: 10.1186/1471-2318-14-91. PMID 25141850
- [Derived] Silva de Lima AL, Hahn T, de Vries NM, Cohen E, Bataille L, Little MA, Baldus H, Bloem BR, Faber MJ. Large-Scale Wearable Sensor Deployment in Parkinson's Patients: The Parkinson@Home Study Protocol. JMIR Res Protoc. 2016 Aug 26;5(3):e172. doi: 10.2196/resprot.5990. PMID 27565186

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After changing the inclusion process for one cohort only, a total of 347 eligible PD patients were invited to participate. Among those invited, 43 refused to participate. The main refusal reasons were "Study protocol seems too burdensome" (44%, n = 19), followed by "Personal circumstances" (33%, n = 14). A total of 304 patients (enrolment rate = 88%) were enrolled.
Groups:
- Cohort 1: Dutch Parkinson's patients who fulfill the eligibility criteria.
  Interventions/Exposures to be administered:
  1. PPMI (Parkinson's Progression Markers Initiative) protocol Trained physiotherapists will perform once a standardized clinical assessment to every included patient. This assessment will last for 60 minutes, and it will be done once.
  2. Fox Insight self-monitoring android app and falls detector Patients will wear a smartwatch and a pendant movement sensor during day and night, for a period of 13 weeks. Additionally, a self-monitoring App on a Smartphone is used, where the patient reports when (s)he takes any PD medication. An additional, optional button allows the patient to report general feeling.
Period: Overall Study
Arm/Group | Cohort 1
Started | 304 (Participants (People with Parkinson's Disease) who signed a consent form.)
Completed | 291 (Participants (People with Parkinson's Disease) who contributed data for 13 weeks.)
Not Completed | 13
Not completed — Withdraw or did not contribute data. | 13

BASELINE CHARACTERISTICS:
Population: Inclusion was changed from 5 cohorts (total of 100 participants) to 1 cohort only.
Arm/Group | Cohort 1
Number analyzed (Participants) | 291
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 261
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123
  Male | 168
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — These data were not reported.
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 0
    Unknown or Not Reported | 291
Disease severity [Count of Participants; unit: Participants] — Participants were assessed using the Hoehn and Yarhn scale. The scale is a grading of the degree of severity of Parkinson's Disease. The scale goes from 0 to 5, in which a higher score indicates higher disease severity.
  Participants
    Stage 0 or 1 | 73
    Stage 2 | 127
    Stage 3 | 34
    Stage 4 or 5 | 6
    Missing | 51
Depression [Count of Participants; unit: Participants] — Depression was assessed using the Geriatric Depression Scale. The total score goes from 0 to 15. A score higher than 6 indicates higher probability of suffer from a depression.
  Participants
    No | 238
    Yes | 53
Cognitive impairment [Count of Participants; unit: Participants] — Cognitive Impairment was measured using the Montreal Cognitive Assessment (MoCA). The MoCA total scores goes from 0 to 30. A score lower than 26 indicates possible presence of Mild Cognitive Impairment.
  Participants
    No | 124
    Yes | 167
Independency level [Number; unit: participants] — Independency Level was assessed using the Modified Schwab and England Activities of Daily Living Scale. The scale goes from 0 to 100. The higher the score, the more independent is the person. We opted for clustering the data into 4 categories because this provided a better overview of participants completely independent, independent, somewhat independent and dependent.
  participants
    Equal or small to 70 | 36
    71-80 | 51
    81-90 | 110
    Equal or higher to 91 | 41
MDS-UPDRS [Median (Full Range); unit: units on a scale] — The Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) was developed to evaluate various aspects of Parkinson's disease, including non-motor and motor experiences of daily living, as well as motor complications. The total score used here was calculated by a sum of all scores from the 4 sub-scales (i.e. part I up to part IV) composing the MDS-UPDRS. Total score ranges from 0 to 272. A higher score indicates higher disease severity and burden, being thus a worse outcome.
  units on a scale | 52.5 [35 to 69]
Age at disease onset. [Mean (Standard Deviation); unit: years] — These data were not reported. Population: Age at disease onset was first included as an outcome. During data-collection, we have chosen not to collect it because other measures (such as MDS-UPDRS) better reflects the impact, burden and severity of the disease.
Time since Diagnose [Mean (Standard Deviation); unit: years] — These data were not reported. Population: Time since diagnose was first included as an outcome. During data-collection, we have chosen not to collect it because other measures (such as MDS-UPDRS) better reflects the impact, burden and severity of the disease.
Level of education [Count of Participants; unit: Participants] — We asked participants to report their highest education finished. After, we categorized answers into: > Highschool - High; < Highschool AND > Middel education - middle; < middel educatoin - low
  Participants
    Low | 51
    Middel | 103
    High | 101
    Missing | 36

OUTCOME MEASURES:

1. Primary Outcome: Parkinson's Disease Symptoms
Description: The MDS-UPDRS is a revision of the Unified Parkinson's Disease Rating Scale (UPDRS). It was developed to evaluate various aspects of Parkinson's disease including non-motor and motor experiences of daily living, as well as motor complications. The MDS-UPDRS characterizes the extent and burden of disease across various populations. Here, we used data from one-point assessment (baseline). The total score used here was calculated by a sum of all scores from the 4 sub-scales (i.e. part I, up to part IV) composing the MDS-UPDRS. Total score ranges from 0 to 272. A higher score indicates higher disease severity and burden, being thus a worse outcome.
Time Frame: Baseline
Population: We have analysed data from all participants who completed the study.
Measure: Median (Full Range); unit: units on a scale
Groups:
- Cohort 1: Dutch Parkinson's patients resident in the region of Noord-Holland whose fulfill the eligibility criteria.
  Interventions/Exposures to be administered:
  1. PPMI (Parkinson's Progression Markers Initiative) protocol Trained physiotherapists will perform once a standardized clinical assessment to every included patient. This assessment will last for 60 minutes, and it will be done once.
  2. Fox Insight self-monitoring android app and falls detector Patients will wear a smartwatch and a pendant movement sensor during day and night, for a period of 13 weeks. Additionally, a self-monitoring App on a Smartphone is used, where the patient reports when (s)he takes any PD medication. An additional, optional button allows the patient to report general feeling.
  Clinical assessment: During the 13 week follow-up, trained physiotherapists will perform a standardized clinical assessment, based on the PPMI protocol (www.ppmi-info.ors) for every included patient. This assessment will last for 60 minutes, and it will be done once.
  Fox Insight self-monitoring android app and falls detector: Patients will be asked to wear a smartwatch and a pendant movement sensor, both with triaxial accelerometers, during day and night, for a period of 13 weeks. Additionally, a self-monitoring App on a Smartphone is used, where the patient reports when (s)he takes any PD medication. An additional, optional button allows the patient to report general feeling.
Arm/Group | Cohort 1
Number analyzed (Participants) | 291
units on a scale | 52.5 [35 to 69]

2. Primary Outcome: Depression Scores as a Measure of Depression Rates
Description: The scores obtained with the Geriatric Depression Scale were analysed in order to create a percentage of probably depressed participants. The total score goes from 0 to 15. A score higher than 6 indicates higher probability of suffer from a depression.
Time Frame: Baseline
Population: We have analyzed all participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 291
Participants
  No | 238
  Yes | 53

3. Primary Outcome: Cognitive Impairment.
Description: Total sum score obtained with the Montreal Cognitive Assessment. We analyzed the full score to investigate percentage of participants with a possible cognitive impairment. The Montreal Cognitive sum scores ranges from 0 to 30, in which a score lower or equal to 26 is considered as possible cognitive decline.
Time Frame: Baseline
Population: We analyzed all participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 291
Participants
  No cognitive decline | 125
  Possible cognitive decline | 166

4. Primary Outcome: Independency Level
Description: The total sum score obtained with the Schwab and England activities of daily living scale were analyzed to describe the functional level of the sample. The total sum scores varies from 0 to 100, in which lower scores are associated with more dependency of others to perform daily life activities.
Time Frame: Baseline
Population: We analyzed all participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 291
Participants
  Lower or equal to 70 | 36
  Higher than 70 and lower than 81 | 51
  Higher than 80 and lower than 91 | 109
  higher than 90 | 41
  Missing | 54

5. Secondary Outcome: Number of Falls Per Patient Registered by the Falls Detector.
Description: The fall event is recognized by the falls detector. Every time that the patient falls, the algorithm embedded at the falls detector recognize as a fall and record the fall event. At the end of the follow-up time, a sum of the falls event for each patient will be done.
Time Frame: Patients will be automatically assessed during the follow-up time (up to 13 weeks after the enrollment date), 24 hours a day, 7 days a week.
Population: We invited 43 study participants to wear the fall detector, of whom 13 consented to wear it. Unfortunately the quality of the collected data did not allow for automated falls detection. Therefore we couldn't determine this outcome measure.
Arm/Group | Cohort 1
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Mood Reports for Each Patient Measured With a Four Point Scale
Description: The number of mood reports will be collected through the smartphone application. A four point scale (very good, good, poor and fair) will be available, and by pressing the button which correspond to how the patient feels at that moment the report can be performed. At the end of the follow-up time a sum of all the reports will be done in order to measure the number of mood reports over the follow-up time.
Time Frame: Patients will be assessed during the follow-up time (up to 13 weeks after the enrollment date). It is expected that the assessment (self-report) will be performed as many times as the patient wants to report how they feel or at least once a day.
Population: Though the smartphone application had to option to report "mood", participants hardly used this feature. Therefore there were no data collection that were suitable for analysis.
Arm/Group | Cohort 1
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Medication Intake Annotations Made by Each Participant Via the Self-report App.
Description: The number of medication intake annotations made by the patients will be collected through the smartphone application. Every time that the patient take medication they must press the button reporting that they took the medication. At the end of the follow-up time a sum of all the reports will be done in order to measure the number of medication intake over the follow-up time.
Time Frame: Baseline
Population: 96% (n = 280) of data-contributors reported their medication through the app.
Measure: Mean (Standard Error); unit: number of annotations
Arm/Group | Cohort 1
Number analyzed (Participants) | 280
number of annotations | 351 (217)

8. Secondary Outcome: Time That Each Patient Was Active During the Day
Description: The time that the patient was active during the day is calculated automatically through the app at the smartphone. The calculation is performed by using an algorithm, which analyze the patterns of walk. This algorithm is able to predict when the patient was active in a zone above his/her usual threshold (e.g. when the patient was performing one activity that makes him/her more active than during a quiet time). At the end of the follow-up time a sum of all active hours will be done in order to measure the amount of time that the patient was active over the follow-up time.
Time Frame: Patients will be automatically assessed continuously during the follow-up time (up to 13 weeks after the enrollment date), 24 hours a day, 7 days a week. The analyses was limited to walking activities.
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Cohort 1
Number analyzed (Participants) | 291
minutes per day | 72 (39)

9. Secondary Outcome: Level of Activity for Each Patient During the Day
Description: The level of activity for each patient is calculated automatically through the app at the smartphone. The calculation is performed by using the data collect with the accelerometers embedded in the smartwatch. An algorithm installed in the phone, which analyze the data collected with the smartwatch, can calculate the level of activity for each patient throughout the day.
Time Frame: as for outcome 5
Population: The collected accelerometer data turned out to be unsuitable to calculate the level of activity during the day. Algorithms produced unreliable information on activity levels and therefore no data on this outcome measure were available.
Arm/Group | Cohort 1
Number analyzed (Participants) | 0

10. Secondary Outcome: Scores in Autonomic Dysfunctions Measure With the Autonomic Dysfunctions Scale
Description: The scores for autonomic dysfunctions will be obtained with the Assessment of autonomic dysfunction in Parkinson's disease (SCOPA-AUT). The total sum scores ranges from 0 to 100, in which high scores are correlated with more burden of autonomic dysfunctions in Parkinson's patients.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1
Number analyzed (Participants) | 245
score on a scale | 17.2 (7.9)

11. Secondary Outcome: Sleepiness Rates in the Epworth Sleepiness Scale as a Measure of Sleep Quantity.
Description: The Epworth sleepiness scale was used to rate the level of sleepiness during the day. The scale's scores are related to the usual duration of sleep at night and increase with relative sleep deprivation. Here, we used data from one-point assessment (baseline). Then, we can suggest that if the sample has high scores they will have a low sleep quantity. Total sum score ranges from 0 (no sleepiness at all) to 24 (excessive sleepiness).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1
Number analyzed (Participants) | 245
score on a scale | 6.0 (4.7)

ADVERSE EVENTS:
Time Frame: 13 weeks
Description: Serious Adverse Events: Include adverse events that result in any of the following outcomes: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect.
  Other (Not Including Serious) Adverse Events: Adverse events that are not Serious Adverse Events.
Groups:
- Cohort 1 (The Study Only Included 1 Cohort).: Dutch Parkinson's patients who fulfill the eligibility criteria.
  Interventions/Exposures to be administered:
  1. PPMI (Parkinson's Progression Markers Initiative) protocol Trained physiotherapists will perform once a standardized clinical assessment to every included patient. This assessment will last for 60 minutes, and it will be done once.
  2. Fox Insight self-monitoring android app and falls detector Patients will wear a smartwatch and a pendant movement sensor during day and night, for a period of 13 weeks. Additionally, a self-monitoring App on a Smartphone is used, where the patient reports when (s)he takes any PD medication. An additional, optional button allows the patient to report general feeling.
Arm/Group | Cohort 1 (The Study Only Included 1 Cohort).
Serious Adverse Events (participants affected / at risk) | 0/291
Other Adverse Events (participants affected / at risk) | 0/291

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes